CLINICAL TRIAL: NCT00600067
Title: A Randomized, Double Blind Multicenter Study to Evaluate the Long-term Safety and Efficacy of VI-0521 Relative to Placebo in Providing and Maintaining Glycemic Control in Type 2 Diabetic Adults
Brief Title: A VI-0521 Study to Evaluate the Long-term Safety and Efficacy in Type 2 Diabetic Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Collaborators: Synteract, Inc. (Industry); Sentrx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DM-230
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes
Keywords: Diabetes; Type 2 Diabetes; Diabetes Mellitus; Metabolic Diseases; Glucose Metabolism Disorders; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Metabolic Diseases; Glucose Metabolism Disorders | interventions — Qsymia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Phentermine/Topiramate
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phentermine/Topiramate — phentermine 15mg/ topiramate controlled release (CR) 92mg, oral capsule, once daily, 28 weeks
  Arms: 1
Drug: Placebo — Oral placebo capsules, once daily, 28 weeks
  Arms: 2

SUMMARY:
The purpose of the study is to determine the long-term safety and efficacy of VI-0521 (phentermine/topiramate) compared to placebo in providing blood sugar control in Type 2 diabetic adults. Continuation of initial 6 month trial.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the qualifying OB-202 trial
* If females of child-bearing potential, subjects must be using adequate contraception
* Provide written informed consent
* Be willing and able to comply with scheduled study visits, treatment plan, lab tests and other study procedures

Exclusion Criteria:

* Subjects who have developed one or more morbidities during the OB-202 trial that would pose a safety concern

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Troupin, MD, MBA, Study Director — VIVUS LLC
Locations (9):
- United States (9):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Spring Valley, California
  - Research Site, Walnut Creek, California
  - Research Site, Bethesda, Maryland
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia

REFERENCES:
- [Derived] Garvey WT, Ryan DH, Bohannon NJ, Kushner RF, Rueger M, Dvorak RV, Troupin B. Weight-loss therapy in type 2 diabetes: effects of phentermine and topiramate extended release. Diabetes Care. 2014 Dec;37(12):3309-16. doi: 10.2337/dc14-0930. Epub 2014 Sep 23. PMID 25249652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment occurred in 10 investigative sites in the U.S. between January 2008 and October 2008
Groups:
- VI-0521: phentermine 15 mg/topiramate 92 mg
Period: Overall Study
Arm/Group | Placebo | VI-0521
Started | 55 | 75
Completed | 52 | 68
Not Completed | 3 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — protocol non-compliance | 0 | 3
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: PHEN/TPM 15/92
- Total: Total of all reporting groups
Arm/Group | Placebo | Active | Total
Number analyzed (Participants) | 55 | 75 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 49.5 (8.58) | 49.7 (7.51) | 49.6 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 58 | 90
  Male | 23 | 17 | 40
Region of Enrollment [Number; unit: participants]
  United States | 55 | 75 | 130

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline Week 0 to Week 56
Time Frame: Baseline to 56 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- VI-0521: phentermine 15mg/topiramate 92 mg
Arm/Group | Placebo | VI-0521
Number analyzed (Participants) | 55 | 75
percent change | -1.2 (0.13) | -1.56 (0.11)
Statistical Analysis 1: Comparison: Placebo vs VI-0521; Test type: Superiority or Other; p = 0.0381, ANCOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.69 to -0.02], Standard Error of Mean 0.17

2. Secondary Outcome: Percent Weight Loss From Baseline to Week 56
Time Frame: Baseline to 56 weeks
Population: Intent-to-treat Last-observation-carried-forward (ITT-LOCF)
Measure: Least Squares Mean (Standard Error); unit: percent change
Groups:
- VI-0521: phentermine 15mg/topiramate 92mg
Arm/Group | Placebo | VI-0521
Number analyzed (Participants) | 55 | 75
percent change | -2.71 (0.95) | -9.41 (0.81)
Statistical Analysis 1: Comparison: Placebo vs VI-0521; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.70, 95% CI 2-sided [-9.18 to -4.21], Standard Error of Mean 1.26

ADVERSE EVENTS:
Time Frame: AEs were collected from when written informed consent was provided through 28 days after the last dose of investigational product.
Arm/Group | Placebo | Active
Serious Adverse Events (participants affected / at risk) | 1/55 | 2/75
Other Adverse Events (participants affected / at risk) | 34/55 | 48/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Active (N=75)
costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Active (N=75)
upper respiratory tract infection (Infections and infestations) | 8 | 7
constipation (Gastrointestinal disorders) | 1 | 4
paresthesia (Nervous system disorders) | 0 | 4
back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
hypoglycemia (Metabolism and nutrition disorders) | 5 | 9
diabetes mellitus (Metabolism and nutrition disorders) | 5 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Influenza (Infections and infestations) | 0 | 2
nasopharyngitis (Infections and infestations) | 1 | 1
bronchitis (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 1 | 1
sinusitis (Infections and infestations) | 1 | 0
diarrhea (Gastrointestinal disorders) | 2 | 0
nausea (Gastrointestinal disorders) | 1 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
abdominal pain (Gastrointestinal disorders) | 1 | 1
dizziness (Nervous system disorders) | 1 | 1
headache (Nervous system disorders) | 1 | 1
hypoesthesia (Nervous system disorders) | 1 | 2
pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
insomnia (Psychiatric disorders) | 0 | 1
anxiety (Psychiatric disorders) | 1 | 0
pyrexia (General disorders) | 2 | 0
vision blurred (Eye disorders) | 2 | 0
hypertension (Vascular disorders) | 1 | 3
depression (Psychiatric disorders) | 0 | 1
hypokalemia (Metabolism and nutrition disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's written notification that publication of results is no longer planned or 12 months after termination of the study at all sites, Institution & PI may publish, upon written approval from Sponsor, results of the Study. Sponsor will be given the opportunity to review any proposed publication at least 60 days prior to submission for publication or disclosure. Upon Sponsor's written request, Institution and PI shall not publish or disclose information related to the Study.